CLINICAL TRIAL: NCT00116025
Title: Pharmacokinetics of Ghrelin in Normal Subjects
Brief Title: Pharmacokinetics of Ghrelin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2004/100; 2004-002207-33; 20040115
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Human acylated ghrelin

SUMMARY:
The main purpose of this study is to determine the half life of the hormone "ghrelin" in the human body. Other purposes are to investigate the effect of ghrelin on appetite and cardiovascular function.

DETAILED DESCRIPTION:
Ghrelin is a recently described acylated peptide hormone produced by the enteroendocrine cells of the mucosal epithelial layer in the ventricle. Ghrelin is the endogenous ligand for the growth hormone (GH) secretagogue receptor (GHS-R).

Ghrelin stimulates pituitary GH release by binding to the GHS-R at both hypothalamic and pituitary levels.

Several studies show that bolus injections of ghrelin have positive effects on cardiac function in healthy humans as well as in humans with cardiac disease. We investigate the changes in cardiac function during ghrelin infusion in healthy subjects.

The pharmacokinetics of ghrelin is described in few studies only, and we aim to elucidate this aspect further.

Comparisons: In a double blind, placebo controlled, cross over study we investigate the effect of 180 minutes ghrelin infusion on 1. cardiac function (tissue Doppler, stroke-velocity index), 2. vascular tone (a. brachialis dilatation), 3. ghrelin-half-life (acylated and des-acylated) and other pharmacokinetic parameters and 4. effect on appetite.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* BMI < 25 kg/m2
* Non-smoker
* Age < 40 yrs

Exclusion Criteria:

* Any known disease
* Any medication (except OTCs)
* Former malignant disease
* Alcoholism
* Blood donation (with in 6 months)
* Allergy to test medication

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17
Dates: Start 2005-03; Study Completion 2006-01

PRIMARY OUTCOMES:
Human ghrelin half life in healthy subjects

SECONDARY OUTCOMES:
Cardiovascular indices (stroke-velocity index, TEI-index)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jorgensen, DrMedSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Vestergaard ET, Gormsen LC, Jessen N, Lund S, Hansen TK, Moller N, Jorgensen JO. Ghrelin infusion in humans induces acute insulin resistance and lipolysis independent of growth hormone signaling. Diabetes. 2008 Dec;57(12):3205-10. doi: 10.2337/db08-0025. Epub 2008 Sep 5. PMID 18776138